CLINICAL TRIAL: NCT01269125
Title: Ultralong Administration of GnRH-a Before in Vitro Fertilization Improves Fertilization Rate But Not Pregnancy Rate in Women With Endometriosis. A Prospective, Randomized, Controlled Trial.
Brief Title: GnRH-a and Pregnancy Rate in In Vitro Fertilization (IVF) Cycles.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Collaborators: University of Patras (Other); Tottori University Hospital (Other)
Responsible Party: Principal Investigator, Apostolos Kaponis, Lecturer of Ob/Gyn, University of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003/89 PGNI
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Endometriosis; Infertility
Keywords: cytokines; endometriosis; fertilization rate; follicular fluid; pregnancy rate
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endometriosis, leuprolide, IVF (Active Comparator): Women with stage II endometriosis received GnRH-a (leuprolide) prior to an IVF attempt.
  Interventions: Drug: Leuprolide; Procedure: IVF
- Endometriosis, IVF (Active Comparator): Women with mild endometriosis who underwent an IVF attempt without prior administration of GnRH-a.
  Interventions: Drug: Leuprolide; Procedure: IVF
- Tubal infertility, IVF (Active Comparator): Women with tubal infertility underwent an IVF attempt.
  Interventions: Procedure: IVF

INTERVENTIONS:
Drug: Leuprolide — single injection of 3.75 leuprolide every 28 days, 3 dosages
  Other Names: Daronda depot 3.75, Abbott, Hellas
  Arms: Endometriosis, IVF; Endometriosis, leuprolide, IVF
Procedure: IVF — Assisted Reproduction Technique.

SUMMARY:
The investigators attempted to establish a rationale for the Gonadotropin Releasing Hormone-agonist (GnRH-a) administration, post-laparoscopically, in women with mild endometriosis (until stage II, according to AFS) who underwent IVF-ET procedure. Since GnRH-a reduces cytokine's concentration in serum (Iwabe et al., 1998; Iwabe et al., 2003) and peritoneal fluid of women with endometriosis (Taketani et al., 1992) the investigators hypothesized that GnRH-a can reduces also cytokine's concentration in the follicular fluid and this action may improve the oocyte quality and the fertility of these women.

DETAILED DESCRIPTION:
This prospective, randomized study with control group was carried out at the Department of Obstetrics and Gynecology, Ioannina University School of Medicine (Ioannina, Greece). The study population consisted of 120 infertile women (more than a year of sexual attempts), aged 29-38 years, with laparoscopically documented endometriosis referred to the In Vitro Fertilization (IVF) Unit of the Department for infertility treatment during a 7-years period (May 2004 to September 2010). In addition, in the current study, we used 60 women with tubal infertility, documented by laparoscopy, without prior history of ovarian surgery, hydrosalpinx, and/or endometriosis as control group. This group was used to see if endometriosis affect the women's fertility. The participant's enrolment was made by three following authors A.K., K.Z., and M.P. During laparoscopy, the endoscopist documented the extension of the disease, the distribution of endometriotic lesions into the peritoneal cavity, and the presence/absence of active endometriotic lesions (red vascularized areas). All visible active endometriotic lesions were cauterized with bipolar diathermy. Women with sonographic evidence of ovarian endometrioma > 2 cm in mean diameter, with early follicular phase serum Follicular Stimulating Hormone (FSH) levels > 12 mIU/ml were excluded from the study. Cases of male factor infertility defined as a concentration of motile sperm less than 10 x 106 /ml and sperm with normal morphology less than 4% (Kruger, strict criteria) were also excluded from the study.

All women who decided to undergo an IVF-Embryo Transfer (ET) attempt were randomized into two groups according to administration or not of GnRH-a treatment, post-laparoscopy. The randomization is performed by accessing a central internet-based randomization program. The random allocation sequence and the assignment of the participants to interventions were made by the first author of the study (A.K.). The first group (Group A) was consisted of 60 women who received a depot preparation of a GnRH-a, 3.75 mg s.c, (leuprolide, Daronda depot, 3.75, Abbott, Hellas) every 28 days for three injections. The investigators preferred to pre-treat study patients with a long-acting GnRH-a for a period of 3 months because it has already reported that pregnancy rates after IVF-ET are similar in patients with endometriosis who are pre-treated with a GnRH-a for 10 to 90 days or greater than 90 days (Caruso 1997; Surrey et al., 2002). In this group, laparoscopies were performed 4 to 6 months prior of any cycle initiation for infertility. The second group (Group B) was consisted of 60 infertile women with endometriosis who did not receive the long-acting GnRH-a. All women were comparable regarding mean age, BMI, and duration of infertility.

All women of control and of group B, underwent controlled ovarian hyperstimulation (COH) after down-regulation with a GnRH-a (leuprolide, 20 IU/day, Daronda, 2.8, Abbott, Hellas) in a long protocol with a mid-luteal start. Administration of recombinant follicle stimulating hormone (rFSH, Gonal-F, Serono, Geneva, Switzeland) was started after at least 14 days of leuprolide therapy and when serum estradiol (E2) had been less than 100 pmol/l and when the thickness of the endometrium was less than 5mm. Down-regulation in women of group A was initiated 30 to 45 days after the third GnRH-a injection. A starting dose of 150 IU of follicle stimulating hormone (rFSH, Gonal-F, Serono, Geneva, Switzerland) was adjusted individually from day 6 of the cycle according to estradiol (E2) values and ultrasonographic follicular measurements. An ovulatory dose of human chorionic gonadotropin (HGG) (Pregnyl, Organon, Oss, The Netherlands) 5,000-10,000 IU was administered I.M. when mean diameter of an average of two to four follicles was larger than 16mm and the plasma estradiol concentration was higher than 1500 pmol/l.

All women were provided to luteal-phase support with natural micronized progesterone (Ultrogestan, Faran, Athens, Greece), 600 mgr daily vaginally in three divided dosages, starting the day after embryos transfer.

Follicular fluid sampling, oocyte collection and IVF Follicular fluid (FF) samples were collected during oocyte retrieval. From each patient, follicular fluid was sampled from the first one to three mature follicles, having a diameter of 18-20mm. Tumor Necrosis Factor(TNF)-a, Interleukine (IL)-1β, IL-6, IL-8 and IL-1-ra were measured in the FF of all women (secondary outcome measures). To prevent any cytokine alterations, only blood-free samples were used. IVF was performed in all cases. The fertilization rates were estimated for every woman 24 hours after oocyte retrieval (primary outcome measure).

Embryo grading and transfer The embryo quality and the clinical pregnancy rate were also primary outcome measures. Embryo development was evaluated 2 days after oocyte pick-up. The number of blastomeres and the proportion of embryo volume occupied by fragments were used for the evaluation. Embryos with < 10%, < 10-20%, < 20-30% and >30% fragments were estimated as grade 1,2,3 and 4, respectively. Three embryos with the highest blastomere number and the best morphology were transferred in each cycle. The remaining high-grade embryos were cryopreserved the same day.

Pregnancy was diagnosed by quantitative β-hCG, two weeks after embryos transfer. Clinical pregnancy was confirmed by observing fetal cardiac activity on transvaginal ultrasound four weeks after a positive pregnancy test. The clinical pregnancy rate and the quality of embryos were estimated in all women. The pregnancy rate was defined as the presence of sonographically visualized cardiac activity per cycle initiated.

ELIGIBILITY:
Inclusion Criteria:

* Infertility
* Mild endometriosis (until stage II)

Exclusion Criteria:

* ovarian endometrioma > 2 cm
* FSH > 12 mIU/ml
* Mail factor infertility

Ages: 29 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2004-05; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Kaponis, MD, Principal Investigator — Ioannina University School of Medicine
Locations (1):
- Dept. of Obstetrics & Gynecology, University Hospital, Ioannina, Epirus, Greece

REFERENCES:
- [Background] Sallam HN, Garcia-Velasco JA, Dias S, Arici A. Long-term pituitary down-regulation before in vitro fertilization (IVF) for women with endometriosis. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004635. doi: 10.1002/14651858.CD004635.pub2. PMID 16437491
- [Background] Rickes D, Nickel I, Kropf S, Kleinstein J. Increased pregnancy rates after ultralong postoperative therapy with gonadotropin-releasing hormone analogs in patients with endometriosis. Fertil Steril. 2002 Oct;78(4):757-62. doi: 10.1016/s0015-0282(02)03338-1. PMID 12372452
- [Background] Fedele L, Parazzini F, Radici E, Bocciolone L, Bianchi S, Bianchi C, Candiani GB. Buserelin acetate versus expectant management in the treatment of infertility associated with minimal or mild endometriosis: a randomized clinical trial. Am J Obstet Gynecol. 1992 May;166(5):1345-50. doi: 10.1016/0002-9378(92)91602-7. PMID 1595789
- [Background] Vercellini P, Crosignani PG, Fadini R, Radici E, Belloni C, Sismondi P. A gonadotrophin-releasing hormone agonist compared with expectant management after conservative surgery for symptomatic endometriosis. Br J Obstet Gynaecol. 1999 Jul;106(7):672-7. doi: 10.1111/j.1471-0528.1999.tb08366.x. PMID 10428523
- [Derived] Kaponis A, Chatzopoulos G, Paschopoulos M, Georgiou I, Paraskevaidis V, Zikopoulos K, Tsiveriotis K, Taniguchi F, Adonakis G, Harada T. Ultralong administration of gonadotropin-releasing hormone agonists before in vitro fertilization improves fertilization rate but not clinical pregnancy rate in women with mild endometriosis: a prospective, randomized, controlled trial. Fertil Steril. 2020 Apr;113(4):828-835. doi: 10.1016/j.fertnstert.2019.12.018. Epub 2020 Mar 5. PMID 32147182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, randomized study with control group was carried out at the Department of Obstetrics and Gynecology, Ioannina University School of Medicine (Ioannina, Greece)during a 7-years period (May 2004 to September 2010).
Pre-assignment Details: Assessed for eligibility (n= 570) Excluded (n= 390)
  * Not meeting inclusion criteria (n= 102)
  * Declined to participate; underwent expectant management or IUI (n= 253)
  * Other reasons; lost to follow up (n=35)
Groups:
- Endometriosis, GnRH-a Treatment, IVF: Women with mild endometriosis who received GnRH-a treatment prior to an IVF attempt.
Period: Overall Study
Arm/Group | Endometriosis, GnRH-a Treatment, IVF | Endometriosis, IVF | Tubal Infertility, IVF
Started | 60 | 60 | 60
Completed | 53 (lost to follow up:4; OHSS: 2; premature luteinization: 1) | 55 (OHSS:4; premature luteinization: 1) | 60
Not Completed | 7 | 5 | 0
Not completed — Adverse Event | 3 | 5 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometriosis, GnRH-a Treatment, IVF | Endometriosis, IVF | Tubal Infertility, IVF | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 60 | 180
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.8 (3.2) | 31.8 (2.1) | 35.4 (1.9) | 33.6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 60 | 180
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy was confirmed by observing fetal cardiac activity on transvaginal ultrasound four weeks after a positive pregnancy test.
Time Frame: June 2004-August 2010
Population: The study period was seven years. Practical issues such as, no more funds for measuring cytokines, my transportation to different University stopped this study before reaching adequate power. The flow of the participants in our Department was low.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Endometriosis, GnRH-a Treatment, IVF | Endometriosis, IVF | Tubal Infertility, IVF
Number analyzed (Participants) | 53 | 55 | 60
percentage | 28.3 [17 to 43] | 25.4 [15 to 39] | 33.3 [17 to 41]
Statistical Analysis 1: Comparison: Endometriosis, GnRH-a Treatment, IVF vs Endometriosis, IVF; Test type: Superiority or Other; p = 0.80, Chi-squared; Odds Ratio (OR) = 0.28, 95% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0

2. Primary Outcome: Embryo Quality (the Percentage of Grade 1 Embryos Per Participant).
Description: Embryo development was evaluated 2 days after oocyte pick-up. The number of blastomeres and the proportion of embryo volume occupied by fragments were used for the evaluation. Embryos with < 10%, < 10-20%, < 20-30% and >30% fragments were estimated as grade 1,2,3 and 4, respectively.
Time Frame: June 2004-August 2010
Measure: Mean (95% Confidence Interval); unit: Percentage of grade 1 embryos
Arm/Group | Endometriosis, GnRH-a Treatment, IVF | Endometriosis, IVF | Tubal Infertility, IVF
Number analyzed (Participants) | 53 | 55 | 60
Percentage of grade 1 embryos | 25.5 [23.25 to 26.94] | 22.6 [20.21 to 33.85] | 27.0 [18.51 to 29.07]

3. Primary Outcome: Fertilization Rate (Percentage of Fertilized Oocytes).
Description: The fertilization rate was estimated for every woman 24 hours after oocyte retrieval
Time Frame: June 2004-August 2010
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Endometriosis, GnRH-a Treatment, IVF | Endometriosis, IVF | Tubal Infertility, IVF
Number analyzed (Participants) | 53 | 55 | 60
percentage | 73.7 [72.90 to 78.87] | 62.7 [57.03 to 66.08] | 75.7 [74.96 to 77.24]

4. Secondary Outcome: Follicular Fluid's TNF-a Concentration.
Description: TNF-a was measured in the FF of all women (secondary outcome measures). To prevent any cytokine alterations, only blood-free samples were used.
Time Frame: June 2004-August 2010
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Endometriosis, GnRH-a Treatment, IVF | Endometriosis, IVF | Tubal Infertility, IVF
Number analyzed (Participants) | 53 | 55 | 60
pg/ml
  TNF-a | 21.4 (6.7) | 38.6 (7.6) | 22.5 (5.4)
  IL-1β | 3.1 (1.1) | 9.3 (4) | 2.9 (0.8)
  IL-6 | 16.7 (5.2) | 32.1 (6.5) | 14.7 (4.4)
  IL-8 | 238.1 (66.4) | 347.8 (59.6) | 241 (46.7)
  IL-1-ra | 166.6 (42.6) | 183 (46) | 151.7 (39.6)

5. Primary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy rate was confirmed by observing fetal cardiac activity on transvaginal ultrasound four weeks after a positive pregnancy test.
Time Frame: 4 weeks after a positive pregnancy test
Population: In order to handle the problem of small sample size bootstrap techniques are used. Ader et al recommend bootstrap procedures(a) distribution is complicated or unknown, (b) a small sample is available. Finally, the bootstrap distribution has been used in order to calculate all the confidence intervals.
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Endometriosis, GnRH-a Treatment, IVF | Endometriosis, IVF | Tubal Infertility, IVF
Number analyzed (Participants) | 53 | 55 | 60
Percentage | 28.3 [17 to 43] | 25.4 [15 to 39] | 33.3 [22 to 47]
Statistical Analysis 1: Comparison: Endometriosis, GnRH-a Treatment, IVF vs Endometriosis, IVF; Test type: Superiority or Other; p = 0.80, Chi-squared; Odds Ratio (OR) = 0.05, 95% CI [-0.2 to 0.3], Standard Error of Mean 0
Statistical Analysis 2: Comparison: Endometriosis, GnRH-a Treatment, IVF vs Tubal Infertility, IVF; In order to handle the problem of small sample size combined with the inability to identify the theoretical statistical distribution of data, bootstrap techniques are used (10). Ader and co-workers recommend the bootstrap procedure when (a) the theoretical distribution is complicated or unknown, and/or (b) power calculations have to be performed and a small sample is available (11). Finally, the bootstrap distribution has been used in order to calculate all the confidence intervals; Test type: Superiority or Other; p = 0.48, Chi-squared; Odds Ratio (OR) = -0.1, 95% CI [-0.4 to 0.2], Standard Error of Mean 0
Statistical Analysis 3: Comparison: Endometriosis, IVF vs Tubal Infertility, IVF; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.22, Chi-squared; Odds Ratio (OR) = -0.15, 95% CI [-0.4 to 0.1], Standard Error of Mean 0

ADVERSE EVENTS:
Time Frame: A 7-year period (2004-2010).
Arm/Group | Endometriosis, GnRH-a Treatment, IVF | Endometriosis, IVF | Tubal Infertility, IVF
Serious Adverse Events (participants affected / at risk) | 2/60 | 4/60 | 0/60
Other Adverse Events (participants affected / at risk) | 1/56 | 1/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometriosis, GnRH-a Treatment, IVF (N=60) | Endometriosis, IVF (N=60) | Tubal Infertility, IVF (N=60)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 2 (2) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.67% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometriosis, GnRH-a Treatment, IVF (N=56) | Endometriosis, IVF (N=60) | Tubal Infertility, IVF (N=60)
Premature luteinization (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes